CLINICAL TRIAL: NCT03854890
Title: Fluorescent Lymphography-Guided Lymphadenectomy Using Indocyanine Green During Laparoscopic Radical Resection Of Rectal Cancer
Brief Title: Fluorescent Lymphography-Guided Lymphadenectomy In Laparoscopic Proctectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, LI XIN-XIANG, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan FLGI
Record Dates: First submitted 2019-02-19; First posted 2019-02-26 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-02

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lymphadenectomy without indocyanine green injection (No Intervention): Laparoscopic lymphadenectomy will be performed in a standard way.
- Lymphadenectomy with indocyanine green injection (Experimental): Injection of indocyanine green to the submucosal layer around rectal cancer 1 day before surgery. Laparoscopic proctectomy with lymph nodes dissection will be performed under near-infrared imaging.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Indocyanine Green will be injected to the submucosal layer around the lesion one day before surgery.
  Arms: Lymphadenectomy with indocyanine green injection

SUMMARY:
The purpose of this study is to compare the number of lymph nodes retrieved with or without the use of intraoperative fluorescence lymphography in laparoscopic radical resection of rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of rectal carcinoma.
* Without multiple primary cancer.
* Without receiving neoadjuvant chemoradiotherapy.
* Sufficient organ function.
* Able to provide written informed consent.

Exclusion Criteria:

* Younger than 18 years or older than 75 years
* Synchronous or metachronous malignancy within 5 years.
* Patients with Intestinal obstruction or perforation or bleeding who require emergency surgery.
* Patients with a history of pelvic irradiation.
* ASA (American Society of Anesthesiologists) grade IV or V.
* Women who are pregnant (confirmed by serum β-Human Chorionic Gonadotropin in women of reproductive age) or breast feeding.
* Severe mental illness.
* Patients with severe emphysema, interstitial pneumonia, or ischemic heart disease who can not tolerate surgery.
* Patients who received steroid therapy within one month.
* Patients or family members misunderstand the conditions and goals of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
The total number of lymph nodes retrieved | During the surgery
The positive number of lymph nodes retrieved | During the surgery

SECONDARY OUTCOMES:
The duration of the operation to remove the lymph nodes | During the surgery
Detection rate of indocyanine green-positive para-aortic lymph node | During the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No